CLINICAL TRIAL: NCT05298592
Title: A Phase 1 First-in-human Study of BMS-986406 as Monotherapy and Combination Therapies in Participants With Advanced Malignant Tumors
Brief Title: A Study of BMS-986406 as Monotherapy and Combination Therapies in Participants With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA111-001; 2021-006872-17 (EudraCT Number); U1111-1270-3670 (Registry Identifier: WHO)
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Advanced Cancer
Keywords: Opdivo®; Immunotherapy
MeSH Terms: interventions — Nivolumab; Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A: BMS-986406 (Monotherapy Dose Escalation) (Experimental)
  Interventions: Biological: BMS-986406
- Part 1B: BMS-986406 + Nivolumab (Combination Dose Escalation) (Experimental)
  Interventions: Biological: BMS-986406; Biological: Nivolumab
- Part 1C: BMS-986406 + Nivolumab (Indication-Specific Dose Expansion) (Experimental)
  Interventions: Biological: BMS-986406; Biological: Nivolumab
- Part 2: BMS-986406 + Nivolumab (Expansion Cohorts) (Experimental)
  Interventions: Biological: BMS-986406; Biological: Nivolumab
- Part 1D: BMS-986406 + Nivolumab + Carboplatin with Pemetrexed or Paclitaxel (Experimental)
  Interventions: Biological: BMS-986406; Biological: Nivolumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Biological: BMS-986406 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Part 1B: BMS-986406 + Nivolumab (Combination Dose Escalation); Part 1C: BMS-986406 + Nivolumab (Indication-Specific Dose Expansion); Part 1D: BMS-986406 + Nivolumab + Carboplatin with Pemetrexed or Paclitaxel; Part 2: BMS-986406 + Nivolumab (Expansion Cohorts)
Drug: Carboplatin — Specified dose on specified days
  Arms: Part 1D: BMS-986406 + Nivolumab + Carboplatin with Pemetrexed or Paclitaxel
Drug: Pemetrexed — Specified dose on specified days
  Arms: Part 1D: BMS-986406 + Nivolumab + Carboplatin with Pemetrexed or Paclitaxel
Drug: Paclitaxel — Specified dose on specified days
  Arms: Part 1D: BMS-986406 + Nivolumab + Carboplatin with Pemetrexed or Paclitaxel

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986406 administered alone, in combination with nivolumab, or in combination with nivolumab and platinum-doublet chemotherapy (PDCT) in participants with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

Parts 1A, 1B, 1C:

* Histologically or cytologically confirmed locally advanced unresectable, metastatic, or recurrent malignant tumor. Eligible tumor types are non-small cell lung cancer (NSCLC), renal cell carcinoma (RCC), pancreatic ductal adenocarcinoma (PDAC), gastric/gastroesophageal junction, castration-resistant prostate cancer (CRPC), ovarian, squamous cell carcinoma of the head and neck (SCCHN), bladder, melanoma, mesothelioma, triple negative breast cancer (TNBC), and soft tissue sarcoma, except for participants with tumors with central nervous system (CNS) metastases as the only site of active disease

Part 1D:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) of non-squamous or squamous histology with Stage IV A/B (as defined by the 8th International Association for the Study of Lung Cancer Classification) or recurrent disease following multi-modal therapy for locally advanced disease, who have not had systemic therapy for metastatic or recurrent disease.

All Parts:

* Measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), Prostate Cancer Working Group 3 (PCWG3) (for prostate cancer), or modified Response Evaluation Criteria in Solid tumors (mRECIST) (for mesothelioma)
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Prior organ or tissue allograft
* Leptomeningeal metastases
* Untreated CNS metastases
* Serious or uncontrolled medical disorders

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 100 days
Number of participants with serious adverse events (SAEs) | Up to 100 days
Number of participants with AEs meeting protocol defined dose-limiting toxicity (DLT) criteria | Up to 28 days
Number of participants with AEs leading to discontinuation | Up to 100 days
Number of participants with death | Up to 100 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 14 days
Time of maximum observed plasma concentration (Tmax) | Up to 14 days
Trough observed plasma concentration (Ctrough) | Up to 14 days
Incidence of anti-drug antibody (ADAs) | Up to 14 days
Objective response rate (ORR) | Up to 24 months
Disease control rate (DCR) | Up to 24 months
Duration of response (DOR) per tumor appropriate criteria: Modified Response Evaluation Criteria in Solid Tumors (mRECIST) for mesothelioma | Up to 24 months
DOR per tumor appropriate criteria: Prostate Cancer Working Group 3 (PCWG3) for prostate cancer | Up to 24 months
DOR per tumor appropriate criteria: Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) for other solid tumor types | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- United States (9):
  - Local Institution - 0021, Birmingham, Alabama
  - University California San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - UCLA Health, Los Angeles, California
  - Local Institution - 0001, Hackensack, New Jersey
  - Carolina BioOncology Institute, PLLC, Huntersville, North Carolina
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Mary Crowley Cancer Research - Medical City Hospital, Dallas, Texas
  - Local Institution - 0006, Richmond, Virginia
- Argentina (4):
  - Local Institution - 0029, Viedma, Río Negro Province
  - Local Institution - 0023, Rosario, Santa Fe Province
  - Local Institution - 0028, Buenos Aires
  - Local Institution - 0032, Córdoba
- Belgium (3):
  - Local Institution - 0018, Jette, Brussels Capital
  - Local Institution - 0015, Edegem, MA
  - Local Institution - 0012, Brussels
- Local Institution - 0031, Kashiwa-shi, Chiba, Japan
- South Korea (4):
  - Local Institution - 0026, Seongnam-si, Gyeonggi-do
  - Local Institution - 0024, Seoul
  - Local Institution - 0027, Seoul
  - Local Institution - 0025, Seoul
- Spain (8):
  - Local Institution - 0008, Málaga, Andaluca
  - Local Institution - 0030, Barcelona
  - Local Institution - 0017, Barcelona
  - Institut Catala dOncologia ICO - Hospital Duran i Reynals Location, Barcelona
  - Local Institution - 0014, Madrid
  - Local Institution - 0009, Madrid
  - Local Institution - 0016, Madrid
  - Local Institution - 0033, Pamplona

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com